CLINICAL TRIAL: NCT04746859
Title: BETTER Women: Community-Based, Primary Care-Linked Peer Health Coaching to Achieve Evidence-Based Preventive Care Goals - A Pragmatic, Wait-List Controlled Effectiveness-Implementation Trial
Brief Title: Evaluation of the Effectiveness and Implementation of the BETTER Women Peer Health Coaching Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Public Health Agency of Canada (PHAC) (Other Government); Women's College Hospital Foundation (Unknown); Women's College Hospital Family Practice Health Centre (Unknown); Barrie and Community Family Health Team (Unknown); University Health Network, Toronto (Other); Applied Health Research Centre (Other); Summerville Family Health Team (Unknown)
Responsible Party: Principal Investigator, Noah Ivers, Clinician-Scientist, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020-0079-E
Record Dates: First submitted 2021-02-04; First posted 2021-02-10 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Chronic Disease; Cancer
Keywords: chronic disease prevention; cancer screening; community health worker; family practice; randomized control trial; hybrid design; process evaluation
MeSH Terms: conditions — Chronic Disease; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients will have a prevention visit with a Prevention Practitioner (a healthcare provider who has received additional training), complete the baseline survey then be invited to receive ongoing support from a trained, volunteer peer health coach, for up to six months. The coach will support the patient as she works towards achieving personalized health goals to reduce her risk of chronic diseases, including cancer. Patients will be administered additional surveys at 3 and 6 months and a final survey at 12 months.
  Interventions: Other: Prevention Visit; Behavioral: Peer health coaching
- Wait-list Control (Other): Patients will have a prevention visit with a Prevention Practitioner (a healthcare provider who has received additional training) and complete a baseline survey, after which they will receive usual care from their healthcare providers. Patients will be administered another survey at 3 months and a final survey at 6 months. After study completion (about 6-months after the initial prevention visit), patients will be invited to receive ongoing support from a trained, volunteer peer health coach, for up to six months. The coach will support the patient as she works towards achieving personalized health goals to reduce her risk of chronic diseases, including cancer.
  Interventions: Other: Prevention Visit

INTERVENTIONS:
Other: Prevention Visit — Patients will have a one-on-one, approximately one-hour long visit with a specially trained Prevention Practitioner. During this visit, they will discuss the patient's health history, their risks for developing chronic diseases, including cancer, and possible steps they can take to reduce those risks. The Prevention Practitioner will also assist the patient to develop and articulate specific goals the patient would like to work on to reduce their risk of chronic diseases.
Behavioral: Peer health coaching — Patients will be invited to register with the software platform used to facilitate peer health coaching. Once they have registered, they will be matched to a peer health coach who will connect with the patient to initiate the process. The coach will work collaboratively with the patient to help her follow through on a step-wise, personalized plan to achieve health goals that were developed with their prevention practitioner. The coach's approach will be informed by principles of brief action planning and motivational interviewing. Coaches will also provide social support, help to navigate to relevant information and community resources, and advise about options for self-monitoring. Coaching will occur over 12-16 sessions via phone calls, text messages, video calls and/or in-person meetings as desired/convenient and in accordance with local public health guidelines.
  Arms: Intervention

SUMMARY:
The Building on Existing Tools To improvE cancer and chronic disease pRevention and screening in primary care (BETTER) Program allows patients in primary care to have a dedicated visit with a prevention practitioner to discuss chronic disease prevention and cancer screening. A prevention practitioner is a health professional, working in primary care, who has received additional training to discuss chronic disease prevention and screening and develop health goals with patients through shared decision-making. Previous studies have shown that this approach increases the number of prevention and screening actions completed by program participants. However, maintenance of health behaviour changes is difficult without on-going support. There is also some evidence that peer-delivered coaching can improve health outcomes in community settings. As such, the BETTER Women program extends the BETTER program by focusing on 40 to 68-year-old women and providing time-limited support for health behaviour change through peer health coaches. Coaches are volunteers - trained in techniques to support health behaviour change - who support women to achieve their health goals over a 6-month period. In this study, the investigators will explore: (i) whether patients who participate in health coaching after a prevention visit are more likely to increase the number of prevention and screening actions that they complete after six months, compared to women who participate in a prevention visit but do not get health coaching; (ii) whether the intervention effects endure six months after the intervention ends; and (iii) the implementation of the program to learn about factors that affect various aspects of the success and sustainability of the program.

DETAILED DESCRIPTION:
While the BETTER program has been shown to successfully increase the number of preventive care and screening actions completed by patient participants after six months, it is known that it is difficult to maintain new health behaviours in the long-term. Unfortunately, it is not feasible to fund health professionals to offer repeated follow-up visits over the time needed to turn initial behaviour changes into long-term habits. Therefore, the investigators are building upon the existing BETTER program by adding a peer health coaching extension that will provide time-limited coaching for patients who want support as they work towards achieving preventive health goals. This approach takes advantage of growing awareness of the role of lay health coaches in improving and extending the quality and value of primary care.

This is a three-site, pragmatic, wait-list-controlled, randomized, Type 1 hybrid effectiveness-implementation trial with blinded outcome collection after 6 months. One site will be an urban, academic, hospital-based clinic; the second will be a clinic serving a greater proportion of patients from rural areas; and the third site will be a suburban clinic with a large South Asian population. Investigators will invite women who are 40-68 years old to have a single visit with a prevention practitioner and receive behaviour change support for up to six months from a health coach. Coaches will do a 24-hr training course, which includes special techniques to support health behaviour change, before they are matched to a patient. At the suburban site, only South Asian peer health coaches will be recruited and this work is being guided by a South Asian Community Advisory Council made up of members of various community organizations in that region. Patients who enroll in BETTER Women will be randomized to receive health coaching either immediately (intervention group) or after a 6-month delay (wait-list control group).

Effectiveness of the program will be assessed by evaluating for each patient, how many of a set of target chronic disease prevention and screening actions were completed at six months, in comparison to baseline. Investigators will also assess whether patients achieved the health goals that they set with their prevention practitioners, physiological markers of health, as well as habits and behaviours related to diet, physical activity, smoking and alcohol use. These outcomes will be collected via electronic surveys administered at baseline, 3- and 6-months* post enrollment as well as through extraction of data from the patients' electronic medical records and BETTER program documents. These outcomes will be compared between the two groups of patients in the study. Additionally, investigators will survey intervention group participants and extract relevant data from their electronic medical records at 12-months* post enrollment.

An embedded process evaluation will be conducted during the trial to examine the implementation of the program. The process evaluation will include collection of program data, electronic surveys administered to patients as well as qualitative interviews with intervention group patients, peer health coaches and prevention practitioners. Investigators will examine how acceptable the program was to patients; whether and why any adaptations were made; how well the program was utilized; how well the coaches delivered the intervention (e.g., what behaviour change techniques were used); how engaged patients and coaches were with the program; and mechanism(s) of action. Ultimately, investigators expect to gain an understanding of the program's sustainability, acceptability, cost-effectiveness, and factors that might impact future attempts at spread and scale.

Investigators expect to see that women in the intervention group (i.e., those who had a health coach) will complete more preventive and screening actions after six months. Investigators also expect to see that women in the intervention group will make more progress on achieving health goals and making lifestyle changes which reduce the risk of chronic diseases and cancers, that the intervention will increase women's access to resources in their primary care clinics and community, as well as improve the women's ability to maintain healthy behaviours.

Note*: The investigators initially planned to collect surveys and data for the primary outcome (for both groups) at 12 months post enrollment. However, due to pandemic-related recruitment challenges, the data collection timeline was amended as described above to allow more time for recruitment within the project timeline.

ELIGIBILITY:
Inclusion Criteria:

* Patient identifies as a woman;
* Patient is 40-68yo;
* Patient has an email address;
* Patient has at least one behavioural risk factor not at target or at least one cancer screening overdue as defined below:

  * Score of less than 9 on the Mediterranean Diet Tool
  * Less than 150 minutes of moderate to vigorous physical activity per week
  * Smoked a cigarette within the last 30 days
  * Average number of drinks per day is ≥1 and/or has >1 drink on any single occasion
  * Due or overdue for one or more of breast, cervical or colorectal cancer screenings;
* Patient has a valid number for the provincial health insurance program (Ontario Health Insurance Program [OHIP]); and
* Patient's medical records for, at least the previous 3 years are accessible through their family physician.

Exclusion Criteria:

* Patient is unable to give informed consent in English due to language, literacy, or competence;
* Patient is unable or unwilling to communicate with the study team to collect outcomes in English via both email and phone; or
* Patient's primary care provider has identified medical comorbidities or other conditions at baseline that might interfere with the patient's ability to follow through on the intervention.

Ages: 40 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Any person who self-identifies as a woman, regardless of sex assigned at birth, and meets all other eligibility criteria will be invited to participate.
Enrollment: 268 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Increased targeted behaviours from baseline | 0, 6 months
  The primary outcome is binary and defined as whether a patient increased the number of completed targeted behaviours from baseline to end of follow-up at 6 months. The targeted behaviours include the status (up to date or out of date) of three cancer screening tests (cervical, breast, colorectal) and the status (meeting evidence-based target or not) of four behavioural determinants for risk of cancer and chronic disease (diet, smoking, alcohol use, physical activity). If a patient meets at least one more target at 6 months than they met at baseline, their outcome will be considered positive.

SECONDARY OUTCOMES:
Goal achievement | 0, 6 months; 12 months for intervention group only
  Percentage of patient-set health goals that was achieved
Breast cancer screening status | 0, 6 months
  Binary assessment of whether the patient is up to date on their breast cancer screening, as per their history and level of risk
Cervical cancer screening status | 0, 6 months
  Binary assessment of whether the patient is up to date on their cervical cancer screening, as per their history and level of risk
Colorectal cancer screening status | 0, 6 months
  Binary assessment of whether the patient is up to date on their colorectal cancer screening, as per their history and level of risk
Diet status | 0, 3, 6 months; 12 months for intervention group only
  Binary assessment of whether the patient's Mediterranean Diet Score is at target (≥9)
Improvement in diet | 0, 3, 6 months; 12 months for intervention group only
  Binary assessment of whether there was an evidence-based improvement (change ≥2) in diet between assessment points
Diet management | 0, 3, 6 months; 12 months for intervention group only
  Binary assessment of whether patient took at least one meaningful action towards diet management
Physical activity status | 0, 3, 6 months; 12 months for intervention group only
  Binary assessment of whether time (in minutes) spent doing moderate to vigorous physical activity in the last seven days is at the evidence-based target (≥150minutes)
Improvement in physical activity | 0, 3, 6 months; 12 months for intervention group only
  Binary assessment of whether or not there was improvement in the physical activity index (PAI) between assessment points
Physical activity management | 0, 3, 6 months; 12 months for intervention group only
  Binary assessment of whether patient took at least one meaningful action towards physical activity management
Smoking status | 0, 3, 6 months; 12 months for intervention group only
  Binary assessment of whether smoking status meets the target of abstinent for the last 30 days
Improvement in smoking | 0, 3, 6 months; 12 months for intervention group only
  Binary assessment of whether the patient's cigarette consumption category, based on consumption of cigarettes per day (cpd), has improved (i.e., cpd decreased) between assessment points
Smoking management | 0, 3, 6 months; 12 months for intervention group only
  Binary assessment of whether patient took at least one meaningful action towards management of smoking behaviour
Alcohol use status | 0, 3, 6 months; 12 months for intervention group only
  Binary assessment of whether alcohol use is at evidence-based target, i.e., number of drinks per day is <1 and never having ≥1 drink on one occasion
Improvement in alcohol use | 0, 3, 6 months; 12 months for intervention group only
  Binary assessment of whether AUDIT risk category has improved (i.e., risk level has decreased) between assessment points
Alcohol use management | 0, 3, 6 months; 12 months for intervention group only
  Binary assessment of whether patient took at least one meaningful action towards management of alcohol use
Up-to-date measurement of glycated haemoglobin (HbA1c) | 0, 6 months; 12 months for intervention group only
  Binary assessment of whether the latest HbA1c measurement is up to date at study end, as per patient's characteristics
HbA1c control | 0, 6 months; 12 months for intervention group only
  Binary assessment of whether the latest measurement, at study end, is up to date and at target (<7%)
HbA1c | 0, 6 months; 12 months for intervention group only
  The most recent and up to date HbA1c measurement for patients with diabetes mellitus (DM)
Glycemic management | 0, 3, 6 months; 12 months for intervention group only
  Binary assessment of whether patient with DM (HbA1c not at target) has taken any meaningful actions towards management of blood sugar through initiation of new antihyperglycemic medication, up-titration of existing antihyperglycemic medications, or discussion with healthcare professional regarding behavioural changes needed to improve blood sugar
Up-to-date measurement of blood pressure (BP) | 0, 6 months; 12 months for intervention group only
  Binary assessment of whether the latest BP measurement is up to date, as per patient's characteristics
BP control | 0, 6 months; 12 months for intervention group only
  Binary assessment of whether the most recent measurement is up to date and at target as per patient's characteristics
Systolic BP | 0, 6 months; 12 months for intervention group only
  The most recent and up to date systolic BP measurement
Diastolic BP | 0, 6 months; 12 months for intervention group only
  The most recent and up to date diastolic BP measurement
Hypertension management | 0, 3, 6 months; 12 months for intervention group only
  Binary assessment of whether patient with BP not at target has taken at least one action towards management of hypertension through initiation of new blood pressure medication, up-titration of existing blood pressure medication, or discussion with healthcare professional regarding behavioural changes needed to improve blood pressure
Up-to-date assessment of low-density lipoprotein (LDL) cholesterol | 0, 6 months; 12 months for intervention group only
  Binary assessment of whether the latest LDL measurement is up to date, as per patient's characteristics
LDL control | 0, 6 months; 12 months for intervention group only
  Binary assessment of whether the most recent LDL measurement is up to date and at target as per patient's characteristics
LDL | 0, 6 months; 12 months for intervention group only
  The most recent and up to date LDL measurement
LDL cholesterol management | 0, 3, 6 months; 12 months for intervention group only
  Binary assessment of whether patient with LDL not at target has taken at least one action towards management of LDL through initiation of new LDL medication, up-titration of existing LDL medication, or discussion with healthcare professional regarding behavioural changes needed to improve cholesterol
Up-to-date assessment for obesity | 0, 6 months; 12 months for intervention group only
  Binary assessment of whether body mass index (BMI) calculation or waist circumference (WC) measurement is up to date, as per patient's characteristics
BMI control | 0, 6 months; 12 months for intervention group only
  Binary assessment of whether latest, up to date BMI is within target (≤ 30kg/m2)
Management of obesity | 0, 3, 6 months; 12 months for intervention group only
  Binary assessment of whether patient with BMI not at target took any meaningful actions towards management of obesity through use of medication or discussion with healthcare professional regarding behavioural changes needed to manage obesity

OTHER OUTCOMES:
Cardiovascular risk | 0, 6 months; 12 months for intervention group only
  10-year cardiovascular risk
Health-related quality of life | 0, 3, 6 months; 12 months for intervention group only
  Health utility score based on European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) health state
Quality-adjusted life year (QALY) | 0, 3, 6 months; 12 months for intervention group only
  An estimation of the combined health utility values derived from responses from EQ-5D-5L and length of life experienced by patient, between measurement time points
Outpatient visits | 6 months
  Number of times patient accessed publicly funded outpatient healthcare services (e.g., visit to primary care physician, outpatient hospital-based services) while enrolled in the study
Emergency room (ER) visits | 6 months
  Number of times patient accessed publicly funded healthcare services from a hospital emergency room while enrolled in the study
Total healthcare costs | 6 months
  The total cost of publicly funded healthcare utilization (outside of delivery of the intervention) by patient while enrolled in the study
Intervention cost/patient | 4 years
  Incremental cost of the intervention (i.e., delivery of peer health coaching only) per patient
Duration of intervention effect | 6, 12 months
  This outcome is ordinal and calculated *only for intervention group patients*. It represents the nature of the change in the number of completed targeted behaviours from end of intervention (at 6 months) to end of follow-up (at 12 months). The targeted behaviours include the status (meeting evidence-based target or not) of four behavioural determinants for risk of cancer and chronic disease (diet, smoking, alcohol use, physical activity). If a patient meets more targets at 12 months compared to 6 months, the patient will be said to have improved. If the same number of targets are met, the patient will be said to be unchanged. If fewer targets are met, the patient will be said to have worsened.

CONTACTS AND LOCATIONS:
Overall Officials: Noah M Ivers, MD, PhD, Principal Investigator — Women's College Hospital; Aisha Lofters, MD, PhD, Principal Investigator — Women's College Hospital
Locations (3):
- Canada (3):
  - Barrie and Community Family Health Team, Barrie, Ontario
  - Summerville Family Health Team, Mississauga, Ontario
  - Women's College Hospital Family Practice Health Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be available for analysis. Data will be shared through secure platforms compliant with PHIPA. Researchers must submit a data access request, including their research proposal, analysis plan, and research ethics board approval.
  Types of Data Available: Baseline and follow-up (3-, 6-, and 12-month) surveys, BETTER Health Survey, Prevention Prescription and Goals, and relevant outcomes from electronic medical records.
  Other Available Documents: Protocol, Survey Instruments, Interview guides
  Applicable Analyses: Health outcomes and behavior change; Economic evaluations; Implementation and process evaluations; Exploratory analyses on effect modifiers and mechanisms of action; Comparative studies on intervention efficacy
  Privacy and Confidentiality: All data will be de-identified to protect participant privacy. Data transfer and storage will comply with PHIPA. Data will be securely stored in a database with access limited to authorized personnel.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available starting from the completion of the primary outcome analysis and will remain available for at least 10 years as mandated by WCH data storage policies.
Access Criteria: External researchers who have a legitimate interest in the data, subject to approval, must submit a detailed data access request, including their research proposal, analysis plan, and plan for research ethics board approval.

REFERENCES:
- [Background] Grunfeld E, Manca D, Moineddin R, Thorpe KE, Hoch JS, Campbell-Scherer D, Meaney C, Rogers J, Beca J, Krueger P, Mamdani M; BETTER Trial Investigators. Improving chronic disease prevention and screening in primary care: results of the BETTER pragmatic cluster randomized controlled trial. BMC Fam Pract. 2013 Nov 20;14:175. doi: 10.1186/1471-2296-14-175. PMID 24252125
- [Background] Bodenheimer TS, Smith MD. Primary care: proposed solutions to the physician shortage without training more physicians. Health Aff (Millwood). 2013 Nov;32(11):1881-6. doi: 10.1377/hlthaff.2013.0234. PMID 24191075
- [Derived] Kithulegoda N, Williams C, Senthilmurugan A, Aimola S, Atkinson J, Banerjee AT, Bazeghi F, Bender JL, Flynn S, Ghatage L, Goulbourne E, Grunfeld E, Heisey R, Rao A, Sutcliffe K, Lofters A, Ivers NM. Assessing the effectiveness of "BETTER Women", a community-based, primary care-linked peer health coaching programme for chronic disease prevention: protocol for a pragmatic, wait-list controlled, type 1 hybrid effectiveness-implementation trial. BMJ Open. 2024 Jul 24;14(7):e085933. doi: 10.1136/bmjopen-2024-085933. PMID 39053957
- See also: Information about the Alcohol Use Disorders Identification Test (AUDIT) — https://auditscreen.org/
- See also: Mediterranean Diet Toolkit (Nov 2018) by Dietitians of Canada — https://www.dietitians.ca/Advocacy/Toolkits-and-Resources
- See also: The screening tool used to provide the physical activity index (PAI) — https://www.gov.uk/government/publications/general-practice-physical-activity-questionnaire-gppaq